CLINICAL TRIAL: NCT03331471
Title: Effect of Alveolar Recruitment Maneuver on Postoprative Pulmonary Complications in the Elderly With Laparoscopic Surgery
Brief Title: Alveolar Recruitment Maneuver During Pneumoperitoneum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-270
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: ARM group-applying alveolar recruitment maneuver Conventional goup-not applying alveolar recruitment maneuver
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- alveolar recruitment maneuver (Active Comparator): FIO2 0.5, TV 6 ml/kg of ideal body weight, PEEP 5 cmH2O and applying alveolar recruitment maneuver (PEEP 10 cmH2O for 3 breath - PEEP 15 cmH2O for 3 breath and PEEP 20 cmH2O for 10 breath) immediate before and after pneumoperitoneum
  Interventions: Procedure: alveolar recruitment maneuver
- conventional ventilation (Experimental): FIO2 0.5, TV 6 ml/kg of ideal body weight, PEEP 5 cmH2O applying during anesthesia
  Interventions: Procedure: conventional ventilation

INTERVENTIONS:
Procedure: alveolar recruitment maneuver — applying alveolar recruitment maneuver using the anesthesia machine
  Other Names: ARM
  Arms: alveolar recruitment maneuver
Procedure: conventional ventilation — conventional ventilation using the anesthesia machine
  Other Names: conventional
  Arms: conventional ventilation

SUMMARY:
Alveolar recruitment maneuver had been reported of improving arterial oxygenation and pulmonary mechanics and reduce the pulmonary complications. Investigator designed this study for comparision of incidence of pulmonary complications after applying alveolar recruitment maneuver during peumoperitoenum for laparoscopic surgery.

DETAILED DESCRIPTION:
Peumopritoneum might increase the pulmonary dead space and deteriorate the pulmonary mechanics. Especially in the eldery, decreased pulmonary function might aggravate negative response to pneumoperitoneum. Alveolar recruitment maneuver had been reported of improving arterial oxygenation and pulmonary mechanics. Investigator designed this study for comparision of the incidences of pulmonary complications after applying alveolar recruitment maneuver or not during peumoperitoenum for laparoscopic surgery in the elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years, patients who undergoing elective laparoscopoic colorectal surgery for cancer under general anesthesia. ASA pysical status I or II

Exclusion Criteria:uncontrolled cardiovascular disease, obstructive pulmonary disorder, acute or chronic inflammatory lesion in lung.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
lung complications | 2 days after laparoscopic surgery
  Incidence of lung complications

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Cheon Lee, Study Chair — Gachon University Gil Medical Center
Locations (2):
- South Korea (2):
  - Gachon University Gil Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon

IPD SHARING:
Plan to Share IPD: No
not yet decided